CLINICAL TRIAL: NCT04133987
Title: Phase II, Randomized, Double-blind, Clinical Tial of the Safety and Immunogenicity of a Tetravalent Dengue Virus Vaccine Admixture TV005 in the Elderly Aged 50-70 Years in Taiwan
Brief Title: Clinical Trial of the Safety and Immunogenicity of a Tetravalent Dengue Virus Vaccine Admixture TV005 in the Elderly Aged 50-70 Years in Taiwan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Centers for Disease Control, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201712180MSD
Record Dates: First submitted 2019-09-23; First posted 2019-10-21 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Dengue
Keywords: tetravalent dengue vaccine; Phase II clinical trial
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tetravalent live attenuated dengue vaccine admixture TV005 (Experimental): Tetravalent live attenuated dengue vaccine admixture TV005
  Interventions: Biological: Tetravalent live attenuated dengue vaccine admixture TV005
- placebo (Placebo Comparator): Plasma-Lyte A
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Tetravalent live attenuated dengue vaccine admixture TV005 — The admixtures of the candidate vaccines each contain 4 live attenuated dengue viruses, each of a different serotype.
  Arms: Tetravalent live attenuated dengue vaccine admixture TV005
Biological: Placebo — PLASMA-LYTE A Injection pH 7.4 (Multiple Electrolytes Injection, Type 1, USP) is a sterile, nonpyrogenic isotonic solution in a single dose container for intravenous administration.
  Arms: placebo

SUMMARY:
Phase II, randomized, double-blind, placebo-controlled study of the safety and immunogenicity of the recombinant live attenuated tetravalent dengue virus vaccine admixture TV005 in the elderly in Taiwan

DETAILED DESCRIPTION:
In Taiwan, people who aged 50 to 70 years accounted for over 40% among those who infected by dengue virus every year. Therefore, to understanding the immunogenicity and safety of TV005 vaccine among people aged 50 to 70 years is important for whether TV005 can be introduced into Taiwan as a major intervention to control dengue. This trial is a phase II, double-blind, multicenter, and placebo-controlled one. The investigators plan to enroll 252 subjects whose age are 50 to 70 years at four study sites. One single-dose TV005 vaccine or placebo will be given subcutaneously. After vaccination, detailed data of the subjective symptoms, physical examination, laboratory examination, and titer of neutralization antibody from all subjects will be recorded. After completion of the present trial, the investigators can clarify the immunogenicity and safety of TV005 among people aged 50 to 70 years.

ELIGIBILITY:
Inclusion Criteria:

1. Man or non-pregnant / non-lactating woman between the ages of 50 years and 70 years at the time of enrollment into the study.
2. Subjects who the investigator believes can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits).
3. Subject who allows to access to their Medical Record.
4. Subjects whose residence is in Taiwan who will remain available for the duration of the study, approximately 3 years following the first vaccination.
5. Good general health as determined by physical examination, laboratory screening, and review of medical history.
6. An informed consent form signed and dated by the subject.
7. If the subject is female, she must be of non-childbearing potential, i.e. surgically sterilized or one year post-menopausal; or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions (i.e. intrauterine contraceptive device; condom and spermicide combination, oral contraceptives or other equivalent hormonal contraception, e.g. progestin implantable, cutaneous hormonal patch or injectable contraceptives) for 30 days prior to vaccination, have a negative pregnancy test prior to vaccination and must agree to continue such precautions for 90 days after completion of the vaccination. For male subject, he must be abstinent or use a condom together with spermicide for 14 days after completion of the vaccination.

Exclusion Criteria:

1. Pregnant or lactating female or female planning to become pregnant within 90 days of receiving an investigational product or planning to discontinue abstinence or contraceptive precautions within 90 days of receiving an investigational product.
2. Acute or chronic, clinically significant neurological, pulmonary, cardiovascular, hepatic, renal, autoimmune, hematologic, endocrine disease or functional defect, as determined by history, physical examination or screening tests that in the opinion of the investigator would, will jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol.
3. Psychiatric, behavioral disorder, or seizures (with the exception of a single febrile seizure in childhood) that in the opinion of the investigator, will affect the ability of the subject to understand and cooperate with the requirements of the study protocol.
4. Self-reported or suspected congenital or acquired immunodeficiency, or asplenia; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroid therapy (prednisone or equivalent, ≥ 0.5 mg/kg/day or 20 mg/day, for more than 2 consecutive weeks within the past 3 months). Inhaled and topical steroids are allowed.
5. HIV infection by screening (by HIV Ag/Ab combo test or HIV Ab test) and confirmatory assays (by Western blot), Hepatitis C virus (HCV) infection by Anti-HCV antibody, or Hepatitis B virus (HBV) infection by Hepatitis B surface antigen (HBsAg) screening or, unwilling to allow HIV, HCV and HBV testing.
6. Screening laboratory values of hemoglobin <9.5 gm/dL in female adults or <11 gm/dL in male adults, neutrophil <1,000 mm3, platelet < 100,000/mm3, Creatinine >1.5 mg/dL, Bilirubin-T >1.5 times of upper limit, or ALT > 2 times of upper limit.
7. History of allergic disease/reaction likely to be exacerbated by any component of the vaccine, or any history of a severe allergic reaction or anaphylaxis.
8. Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures.
9. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol.
10. Planned administration of any vaccine not foreseen by the study protocol, during the period starting from 30 days before the study vaccine and ending 30 days after study vaccination; with the exceptions of the inactivated influenza vaccine or the inactivated rabies vaccine (without administration of immunoglobulin) administered.
11. Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the study vaccine/placebo or planned use at any time during the study period or history of having received any investigational dengue vaccine at any previous time.
12. Administration of immunoglobulins and/or blood products within 90 days preceding the study vaccine dose or planned administration at any time during the study period, which might interfere with assessment of the immune response. Or administration of killed vaccine within 14 days, or attenuated vaccine within 28 days.
13. A planned or anticipated move to a location that will prohibit participating in the trial for the 12-month duration and unavailable for schedule visit during 2nd and 3rd year follow-up.
14. Potential volunteers who do not have easy access to a fixed or mobile telephone.
15. Any subject identified as a site employee of the Investigator or study clinic, with direct involvement in the proposed study or other studies under the direction of that Investigator or study clinic, as well as any family member (i.e., immediate, husband, wife and their children, adopted or natural) of the clinic employees or the Investigator.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of study participants with solicited local and general adverse events. | Measured through Day 21
Proportion of study participants with unsolicited adverse events. | Measured through Day 29
Proportion of study participants with serious adverse events. | Measured through Day 1080
Evaluation of the immunogenicity of TV005, as assessed by PRNT50 to DENV-1, DENV-2, DENV-3, and DENV-4 at 28, 56, 72 and 180 days after TV005 vaccination | Measured through Day 180

SECONDARY OUTCOMES:
Evaluation of the frequency and quantity of viremia of each monovalent component of the vaccine after vaccination. | Measured through Day 21
Number of TV005 vaccinees infected with DENV-1, DENV-2, DENV-3, and DENV-4. | Measured through Day 72

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided